CLINICAL TRIAL: NCT00552279
Title: Immunogenicity and Safety Study of GlaxoSmithKline Biologicals' HPV Vaccine GSK580299 Administered According to an Alternative Dosing Schedule as Compared to the Standard Dosing Schedule in Young Female Subjects Aged 15-25 Years
Brief Title: Immunogenicity and Safety of GlaxoSmithKline Biologicals' Huma Papillomavirus (HPV) Vaccine 580299 in Healthy Females 15 - 25 Years of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 109179
Record Dates: First submitted 2007-10-30; First posted 2007-11-01 (Estimated); Results first posted 2010-03-05 (Estimated); Last update posted 2018-06-25 (Actual); Status verified 2017-04

CONDITIONS: Infections, Papillomavirus
Keywords: HPV; cervical cancer; papillomavirus; Human papillomavirus (HPV) vaccine
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms | interventions — Papillomavirus Vaccines

ARMS (2):
- Cervarix-12 Group (Experimental): Women received 3 doses of Cervarix TM (human papillomavirus (HPV) vaccine) administered according to a 0, 1, 12-month schedule
  Interventions: Biological: Cervarix TM
- Cervarix-6 Group (Active Comparator): Women received 3 doses of Cervarix TM (HPV vaccine) administered according to a 0, 1, 6-month schedule.
  Interventions: Biological: Cervarix TM

INTERVENTIONS:
Biological: Cervarix TM — Intramuscular administration into the deltoid region of the non-dominant arm according to a 0, 1, 12-month schedule.
  Other Names: HPV vaccine (GSK580299)
  Arms: Cervarix-12 Group
Biological: Cervarix TM — Intramuscular administration into the deltoid region of the non-dominant arm according to a 0, 1, 6-month schedule.
  Arms: Cervarix-6 Group

SUMMARY:
Infection with human papillomavirus (HPV) has been clearly established as the central cause of cervical cancer. The current phase 3b study is designed to assess the immunogenicity and safety of GlaxoSmithKline Biologicals' HPV vaccine GSK580299 administered according to an alternative dosing schedule as compared to the standard dosing schedule in young female subjects aged 15 - 25 years. The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they and/or their parent(s)/Legally acceptable representative(s) (LAR) can and will comply with the requirements of the protocol
* A female between and including 15 and 25 years of age at the time of the first vaccination.
* Written informed consent obtained from the subject prior to enrolment. For subjects below the legal age of consent, written informed consent must be obtained from the subject's parents/legally acceptable representative (LAR), and written informed assent must be obtained from the subject.
* Healthy subjects as established by medical history and/or clinical examination before entering into the study.
* Subject must be of non-childbearing potential, or if she is of child bearing potential, she must practice adequate contraception for 30 days prior to vaccination, have a negative urine pregnancy test and continue such precautions for 2 months after completion of the vaccination series.
* Subject who had no more than 6 lifetime sexual partners prior to enrolment.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Planned administration/administration of a vaccine not foreseen by the study protocol within 30 days before and 30 days after the first dose of vaccine. Planned administration/administration of routine vaccines up to 8 days before the first dose of study vaccine is allowed. Enrolment will be deferred until the patient is outside of specified window.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* Previous vaccination against HPV or planned administration of any HPV vaccine other than that foreseen by the study protocol during the study period.
* previous administration of components of the investigational vaccine
* Cancer or autoimmune disease under treatment.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Hypersensitivity to latex
* Acute disease at the time of enrolment.
* Administration of immunoglobulins and/or any blood products within the three months preceding blood sampling.
* Pregnant or breastfeeding female.
* Female planning to become pregnant, likely to become pregnant (as determined by the investigator) or planning to discontinue contraceptive precautions during the study period starting at visit one and up to two months after the last vaccine dose.
* Acute or chronic clinically significant pulmonary, cardiovascular, hepatic or renal function abnormality as determined by physical examination or lab tests.

Ages: 15 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 805 (Actual)
Dates: Start 2007-11-12; Primary Completion 2009-02-26 (Actual); Study Completion 2009-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (13):
- Italy (7):
  - GSK Investigational Site, Brescia, Lombardy
  - GSK Investigational Site, Lodi, Lombardy
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Cagliari, Sardinia
  - GSK Investigational Site, Sassari, Sardinia
  - GSK Investigational Site, Palermo, Sicily
  - GSK Investigational Site, Ragusa, Sicily
- Romania (3):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Cluj-Napoca
  - GSK Investigational Site, Sibiu
- Slovakia (3):
  - GSK Investigational Site, Dolný Kubín
  - GSK Investigational Site, Nová Dubnica
  - GSK Investigational Site, Trenčín

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Esposito S, Birlutiu V, Jarcuska P, Perino A, Man SC, Vladareanu R, Meric D, Dobbelaere K, Thomas F, Descamps D. Immunogenicity and safety of human papillomavirus-16/18 AS04-adjuvanted vaccine administered according to an alternative dosing schedule compared with the standard dosing schedule in healthy women aged 15 to 25 years: results from a randomized study. Pediatr Infect Dis J. 2011 Mar;30(3):e49-55. doi: 10.1097/INF.0b013e318206c26e. PMID 21273939
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 109179 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 109179 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 109179 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 109179 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 109179 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 109179 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 109179 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 805 subjects were enrolled and 804 subjects were vaccinated and included in the analyses.
Groups:
- Cervarix-12 Group: Women received 3 doses of Cervarix™ (human papillomavirus [HPV] vaccine) administered according to a 0, 1, 12-month schedule.
- Cervarix-6 Group: Women received 3 doses of Cervarix™ (HPV vaccine) administered according to a 0, 1, 6-month schedule.
Period: Overall Study
Arm/Group | Cervarix-12 Group | Cervarix-6 Group
Started | 403 | 401
Completed | 389 | 398
Not Completed | 14 | 3
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 12 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Other | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cervarix-12 Group | Cervarix-6 Group | Total
Number analyzed (Participants) | 403 | 401 | 804
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.6 (2.98) | 18.7 (3.13) | 18.6 (3.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 403 | 401 | 804
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Seroconverted for Anti-human Papilloma Virus 16 (Anti-HPV-16) and Anti-human Papilloma Virus 18 (Anti-HPV-18) Antibodies
Description: Seroconversion is defined as the appearance of anti-HPV-16 and/or anti- HPV-18 antibodies (i.e. antibody titer ≥ cut-off value) in the sera of subjects seronegative before vaccination.
  Cut-off values were 8 enzyme-linked immunosorbent assay units per milliliter (EL.U/mL) for anti-HPV-16 antibodies and 7 EL.U/mL for anti- HPV-18 antibodies.
Time Frame: One month after the third vaccine dose
Population: Analysis was performed on initially seronegative subjects from the According-to-Protocol (ATP) cohort for analysis of immunogenicity
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix-12 Group | Cervarix-6 Group
Number analyzed (Participants) | 346 | 346
Participants
  Anti-HPV-16: number analyzed (Participants) | 337 | 342
  Anti-HPV-16 | 337 | 342
  Anti-HPV-18 | 345 | 346

2. Primary Outcome: Titer of Anti-HPV-16 and Anti-HPV-18 Antibodies
Description: Titer given as geometric mean titer (GMT).
Time Frame: One month after the third vaccine dose
Population: Analysis was performed on initially seronegative subjects from the ATP cohort for analysis of immunogenicity
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Cervarix-12 Group | Cervarix-6 Group
Number analyzed (Participants) | 346 | 346
EL.U/mL
  Anti-HPV-16: number analyzed (Participants) | 337 | 342
  Anti-HPV-16 | 11337.2 [10238.2 to 12554.1] | 10050.9 [9180.9 to 11003.3]
  Anti-HPV-18 | 4526.7 [4110.1 to 4985.6] | 3879.9 [3532.7 to 4261.2]

3. Secondary Outcome: Number of Subjects Seroconverted for Anti-HPV-16 and Anti-HPV-18 Antibodies
Description: as for outcome 1
Time Frame: One month after the second vaccine dose
Population: Analysis was performed on initially seronegative subjects from the ATP cohort for analysis of immunogenicity
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix-12 Group | Cervarix-6 Group
Number analyzed (Participants) | 346 | 346
Participants
  Anti-HPV-16: number analyzed (Participants) | 337 | 342
  Anti-HPV-16 | 337 | 342
  Anti-HPV-18 | 346 | 346

4. Secondary Outcome: Titer of Anti-HPV-16 and Anti-HPV-18 Antibodies
Description: Titer given as GMT.
Time Frame: One month after the second vaccine dose
Population: Analysis was performed on initially seronegative subjects from the ATP cohort for analysis of immunogenicity
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Cervarix-12 Group | Cervarix-6 Group
Number analyzed (Participants) | 346 | 346
EL.U/mL
  Anti-HPV-16: number analyzed (Participants) | 337 | 342
  Anti-HPV-16 | 3307.0 [3051.0 to 3584.5] | 3184.1 [2938.3 to 3450.5]
  Anti-HPV-18 | 2382.3 [2179.2 to 2604.3] | 2256.3 [2070.7 to 2458.7]

5. Secondary Outcome: Number of Subjects Reporting Solicited Local Symptoms
Description: Solicited local symptoms assessed include pain, redness and swelling at the injection site.
Time Frame: During the 7-day (Days 0-6) period following each vaccination
Population: Analysis was performed on the Total Vaccinated Cohort, on subjects with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix-12 Group | Cervarix-6 Group
Number analyzed (Participants) | 402 | 401
Participants
  Pain | 385 | 386
  Redness | 201 | 182
  Swelling | 158 | 145

6. Secondary Outcome: Number of Subjects Reporting Solicited General Symptoms
Description: Solicited general symptoms assessed include arthralgia, fatigue, fever, gastrointestinal symptoms, headache, myalgia, rash, and urticaria.
Time Frame: During the 7-day (Days 0-6) period following each vaccination
Population: Analysis was performed on the Total Vaccinated Cohort, on subjects with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix-12 Group | Cervarix-6 Group
Number analyzed (Participants) | 402 | 401
Participants
  Arthralgia | 85 | 78
  Fatigue | 245 | 237
  Temperature ≥ 37.5°C | 37 | 29
  Gastro-intestinal symptoms | 85 | 86
  Headache | 203 | 199
  Myalgia | 167 | 168
  Rash | 30 | 34
  Urticaria | 12 | 18

7. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AE)
Description: An AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: During the 30-day (Days 0-29) period following each vaccination
Population: Analysis was performed on the Total Vaccinated Cohort, on subjects with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix-12 Group | Cervarix-6 Group
Number analyzed (Participants) | 403 | 401
Participants | 117 | 129

8. Secondary Outcome: Number of Subjects Reporting New Onset of Chronic Diseases (NOCDs), New Onset Autoimmune Diseases (NOADs), Serious Adverse Events (SAEs), and Medically Significant Conditions (MSCs)
Description: Entire study period = up to Month 18 Cervarix-12 & Month 12 Cervarix-6.
  NOCDs assessed include eg. autoimmune disorders (NOADs), asthma, type I diabetes. MSCs assessed include AEs prompting emergency room visits and physician office visits not related to common illnesses.
  An SAE is any untoward medical occurrence that: results in death, is lifethreatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study subject, or may evolve into one of the outcomes listed above.
Time Frame: During the entire study period (up to Month 18 or up to Month 12)
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix-12 Group | Cervarix-6 Group
Number analyzed (Participants) | 403 | 401
Participants
  MSCs | 42 | 44
  NOCDs | 0 | 5
  NOADs | 0 | 2
  SAEs | 12 | 9

9. Secondary Outcome: Number of Subjects With Pregnancies and Their Outcomes
Description: Entire study period = up to Month 18 Cervarix-12 & Month 12 Cervarix-6
  Number of pregnancies and pregnancy outcomes.
Time Frame: During the entire study period (up to Month 18 or Month 12)
Population: Analysis was performed on the Total vaccinated cohort, on pregnant subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix-12 Group | Cervarix-6 Group
Number analyzed (Participants) | 5 | 3
Participants
  Normal infant | 2 | 1
  Elective abortion | 0 | 2
  Abortion threatened | 1 | 0
  Ongoing | 1 | 0
  Foetal distress syndrome | 1 | 0

10. Secondary Outcome: Number of Subjects Completing the 3-dose Vaccination Schedule
Time Frame: After the third vaccine dose
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix-12 Group | Cervarix-6 Group
Number analyzed (Participants) | 403 | 401
Participants | 388 | 397

ADVERSE EVENTS:
Description: Analysis for other adverse events were performed on the Total vaccinated cohort, on subjects with available data.
Arm/Group | Cervarix-12 Group | Cervarix-6 Group
Serious Adverse Events (participants affected / at risk) | 12/403 | 9/401
Other Adverse Events (participants affected / at risk) | 388/403 | 389/401
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cervarix-12 Group (N=403) | Cervarix-6 Group (N=401)
Appendicitis (Infections and infestations) | 2 | 1
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Cyst (General disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Tendon injury (Injury, poisoning and procedural complications) | 1 | 0
Thyroiditis (Endocrine disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Tracheitis (Infections and infestations) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Brain hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cephalhaematoma (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Foetal distress syndrome (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cervarix-12 Group (N=403) | Cervarix-6 Group (N=401)
Pain (General disorders) | 385 | 386
Redness (General disorders) | 201 | 182
Swelling (General disorders) | 158 | 145
Arthralgia (General disorders) | 85 | 78
Fatigue (General disorders) | 245 | 237
Temperature ≥ 37.5°C (General disorders) | 37 | 29
Gastrointestinal symptoms (General disorders) | 85 | 86
Headache (General disorders) | 203 | 199
Myalgia (General disorders) | 167 | 168
Rash (General disorders) | 30 | 34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.